CLINICAL TRIAL: NCT03487458
Title: Quality of Life in Patients With Traumatic Rib Fracture After Rib Fracture Surgery: A Prospective Cohort Study
Brief Title: Quality of Life in Patients With Traumatic Rib Fracture After Rib Fracture Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201703114RIND
Record Dates: First submitted 2017-11-05; First posted 2018-04-04 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2017-06

CONDITIONS: Rib Fractures
MeSH Terms: conditions — Rib Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): participants receive no surgical treatment
- Rib Fixation Surgery (Experimental): participants receive surgical treatment
  Interventions: Procedure: Rib Fixation Surgery

INTERVENTIONS:
Procedure: Rib Fixation Surgery — Rib Fixation Surgery
  Arms: Rib Fixation Surgery

SUMMARY:
This study is a prospective study. Patients with traumatic rib fractures are divided into control group and surgical (OP) group, depending on whether they undergo rib fracture fixation surgeries. They complete Short Form-36 and Work Quality Index (WQI) before surgery and after surgery (before discharge, post-surgery 1 month, 3 months and 6 months). The goal of this study is to examine the life quality of patients who receive surgical treatment for rib fracture by analyzing patients' response, comorbidity, vital signs (blood pressure, heart rate, respiratory rate, Glasgow Coma Scale (GCS) etc.), severity of fracture (AIS, ISS) and medical costs. The investigators hope to find the most suitable method of treatment for patients with rib fractures.

DETAILED DESCRIPTION:
Traumatic rib fracture is one of the most common thoracic traumas. Patients often complain of severe pain of the fracture site, especially when coughing, sneezing, inhaling and lifting arms. If there is obvious displacement of the rib fracture, there are risks of life-threatening open pneumothorax, hemothorax and internal bleeding. Multiple rib fractures may even cause flail chest, leading to respiratory distress and respiratory failure.

Even patients with mild rib fractures may suffer from pain, causing movement limitations and poor sleep. Those whose occupations require heavy labors may even lose their jobs.

Large wounds and difficulties with localization and fixation made surgical interventions a poor option in the past. Thus, treatment goals were set on pain control and infection prevention. However, in recent years, there are improvements with medical imaging, endoscopy and fracture fixation instruments, so rib fracture fixations become a new treatment option. In addition, patients now ask for higher life quality after the trauma recovery, and not just passively controlling the pain and infection.

Therefore, this study is a prospective study. The investigators enrolled patients with traumatic rib fractures from the National Taiwan University Hospital and Far Eastern Memorial Hospital from July 2017 to July 2018. This study incorporated the use of Short Form-36 and Work Quality Index (WQI) to compare the control groups and the surgical (OP) groups. The participants would complete the questionnaires before surgery and after surgery (before discharge, post-surgery 1 month, 3 months and 6 months).

The goal of this study is to examine the life quality of patients who receive surgical treatment for rib fracture by analyzing patients' response, comorbidity, vital signs (blood pressure, heart rate, respiratory rate, GCS etc.), severity of fracture (AIS, ISS) and medical costs. The investigators hope to find the most suitable method of treatment for patients with rib fractures.

ELIGIBILITY:
Inclusion Criteria:

Absolute Indications:

1. Flail chest with paradoxical respiration
2. Multiple rib fractures with uncontrolled hemothorax or pneumothorax
3. Severe thoracic trauma causing respiratory failure (ex poor blood oxygen saturation, hypercapnia, overtime intubation etc.)

Relative Indications:

1. Fractures of 3 or more ribs, with moderate amount of hemothorax or pneumothorax
2. Fractures of 3 or more ribs, with clavicle or scapula fractures, requiring surgical intervention
3. Fractures of 3 or more ribs, with obvious rib displacement and pain
4. Chronic neuropathic pain, with poor drug control
5. Symptoms due to poor healing of fracture site (ex. dyspnea or restrictive lung disease)
6. Chest deformity or other cosmetic factors
7. Other personal factors (ex. disability caused by rib fractures)

Exclusion Criteria:

1. High risk for surgery (ex. Age greater than 75 y/o, poor cardiopulmonary function, abnormal coagulation, end-stage renal disease, hepatic failure etc.)
2. Severe chest trauma, with large area of lung contusion or pulmonary embolism
3. More than 2 organs of systemic severe trauma (ex. combining head trauma, abdominal internal bleeding, abdominal organ rupture etc.)
4. Poor rib fracture site (ex. posterior axillary line, 1st-3rd rib, sub-scapula etc.)
5. Patient refuses surgery
6. current acute infection
7. Allergy to surgical instruments
8. Lack of sufficient blood supply, poor bone density or potential infection
9. Psychiatric or neuropathic conditions causing inability to obey doctor's order

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-06-13 (Actual); Primary Completion 2018-06-12 (Estimated); Study Completion 2018-06-12 (Estimated)

PRIMARY OUTCOMES:
Short Form-36 (SF-36) | Assessment of change in SF-36 scores for the control group at admission and after discharge for up to six months and for the surgical group before and after surgery for up to 6 months.
  questionnaire filled by patient

SECONDARY OUTCOMES:
Work Quality Index (WQI) | Assessment of change in WQI for the control group at admission and after discharge for up to six months and for the surgical group before and after surgery through study completion for up to 6 months.
  questionnaire filled by patient
Days of admission | Assessment of total number of days of hospitalization including ICU stay after admission through study completion for up to 6 months.
  Days of admission in the hospital
Severity of hemothorax | Assessment of progression or resolution of hemothorax after simple chest drainage for up to 3 days after chest drainage insertion in the control group and before operation, post-OP day 1, and post-OP day 3 for up to 3 days' post-operation in the surgical
  The severity of hemothorax is evaluated by amount of chest tube drainage measured in milliliters per day.
Pain | Every 8 hours during hospitalization for up to 1 month and outpatient follow-up at 1 month, 3 months and 6 months after discharge through study completion for a total of 6 months.
  The Numeric Rating Scale (NRS-11), with a scale from 0 to 10, with 0 as no pain, 10 as extremely painful

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan